CLINICAL TRIAL: NCT01379066
Title: Detection of Mycobacteria in Lungs and Culture Using an Ultra-fast Gas Chromatograph
Brief Title: Tuberculosis Volatile Organic Compounds
Acronym: TBVOC
Status: Completed | Type: Observational
Sponsor: Landon Pediatric Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TB1
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Pulmonary Tuberculosis
Keywords: Mycobacterium tuberculosis; Pulmonary tuberculosis; Electronic nose; Gas chromatography
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tuberculosis Patients: Suspected Tuberculosis patients
- Control: Healthy volunteers

SUMMARY:
The Pulmonary Colonization Test is a non-invasive breath test for markers of lower respiratory tract infection, which may predict the probability of mycobacterial organisms in the lower respiratory tract. It consists of:

* A breath collection apparatus for collection of volatile organic compounds in breath onto a sorbent trap and Tedlar bag, as well as for the collection of a separate sample of room air.
* Analysis of the volatile organic compounds in breath and room air by short acoustic wave/gas chromatography.
* Interpretation of the volatile organic compounds with a proprietary algorithm in order to predict the probability of lower respiratory tract colonization and infection.
* Analysis of the volatile organic compounds in sputum culture by short acoustic wave/gas chromatography.

This study will test the hypothesis that the investigators can identify the presence of mycobacteria in an individual by sampling the breath of patients with active tuberculosis and by sampling "head space" above culture media of sputum provided. This study will test the hypotheses:

* that the investigators can identify positive cultures for mycobacterium tuberculosis through sampling of the headspace above the cultures prior to standard laboratory culture identification
* that the investigators can identify control of tuberculosis by sampling exhaled breath

ELIGIBILITY:
Inclusion Criteria:

* Suspected tuberculosis infection or disease
* Positive tuberculosis skin test
* Positive sputum culture for TB
* X-rays indicated possible tuberculosis infection or disease
* ability to give breath and sputum samples at regular intervals

Exclusion Criteria:

* Heavy smoker
* History of or active pulmonary disease other than tuberculosis

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Tuberculosis patients will be enrolled through the Tuberculosis Specialty Clinic in Oxnard, Ca.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Identification of tuberculosis from bacterial plates | 6 months
  Tuberculosis will be identified form culture plates by the volatile organic compound signature

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Oxnard Specialty Clinic, Oxnard, California
  - Pediatric Diagnostic Center, Ventura, California